CLINICAL TRIAL: NCT06391944
Title: A Phase 2, Open Label, Multi-center Study to Assess the Efficacy and Safety of JMT101 Combined With Osimertinib in Patients With Stage Ⅲb-Ⅳ Non-Small Cell Lung Cancer With EGFR Common Mutations
Brief Title: JMT101 Combined With Osimertinib in Patients With Stage Ⅲb-Ⅳ Non-small Cell Lung Cancer (NSCLC) Characterized by Epithermal Growth Factor Receptor (EGFR) Common Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-CSP-005
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Local Advanced or Metastatic NSCLC; Harboring EGFR Common Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: For cohort 1, patients received JMT101 6mg/Kg Q3W and Osimertinib 80mg QD. For cohord 2, patients received JMT101 6mg/Kg Q2W and Osimertinib 80mg QD.For cohort 3 and cohort 4, patients were randomized 1:1 to JMT101 6mg/Kg and Osimertinib 80mg or JMT101 6mg/Kg and Osimertinib 160mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JMT101 combined with Osimertinib (Experimental): JMT101 6mg/kg iv Q2W or Q3W, osimertinib 80mg or 160mg po QD until a treatment discontinuation criterion is met.
  Interventions: Drug: JMT101 Injection; Drug: Osimertinib tablet

INTERVENTIONS:
Drug: JMT101 Injection — JMT101 Injection, 6 mg/kg intravenously, over 90 mins every 14 or 21 days
Drug: Osimertinib tablet — Osimertinib 80 or 160mg po everyday

SUMMARY:
This was a multicenter, open-label phase 2 study. This study aimed to evaluate the efficacy and safety of JMT101 combined with Osimertinib in participants with local advanced or metastatic non-small-cell lung cancer harbouring EGFR common mutation with or without prior systemic therapy.

Efficacy indexes included investigator-assessed Overall Response Rate(ORR), Disease Control Rate(DCR), Duration of Response( DoR), Progression Free Survival (PFS) per RECIST 1.1 and Overall Survival (OS). Safety indexes included Adverse Events incidence and severity. This study included 4 cohorts, cohort 1 included EGFR-mutated advanced NSCLC patients without prior systemic therapy and accepted JMT101 6mg/Kg Q3W and Osimertinib 80mg QD therapy. Cohort 2 included EGFR-mutated advanced NSCLC patients who failed with prior generation 1 or 2 EGFR-TKIs therapy and accepted JMT101 6mg/Kg Q2W and Osimertinib 80mg QD therapy. Cohort 3 included advanced EGFR common mutation NSCLC patients who failed with prior generation 3 EGFR-TKIs but did not accept chemotherapy and accepted JMT101 6mg/Kg Q2W and Osimertinib 80mg or 160mg QD therapy. Cohort 4 included EGFR-mutated advanced EGFR NSCLC patients who failed with prior generation 3 EGFR-TKIs and platinum-based chemotherapy and accepted JMT101 6mg/Kg Q2W and Osimertinib 80mg or 160mg QD therapy.

DETAILED DESCRIPTION:
Avoid duplicating information that will be entered elsewhere, such as Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old.
2. Histologically or cytologically confirmed diagnosis of NSCLC, locally advanced (Stage IIIB and IIIC according to the 8th edition of the AJCC TNM staging criteria) or metastatic (Stage IV) harbouring EGFR common mutation with tumour tissue/blood sample. For cohort 1, should not receive prior systemic therapy, for cohort 2, should fail with generation 1 or 2 EGFR-TKIs therapy, for cohort 3, should fail with generation 3 EGFR-TKIs therapy but did not accept chemotherapy, for cohort 4, patients should fail with generation 3 and platinum-based chemotherapy.
3. At least 1 measurable lesion per RECIST Version 1.1.
4. Life expectancy ≥ 12 weeks.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Adequate organ and hematologic function
7. Women with fertility tested negative for blood pregnancy within 7 days prior to trial screening; Any male or female patients with fertility must agree to use effective contraceptive methods throughout the entire trial period and within six months after the end of the trial.
8. Patients must give informed consent to this study before the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Previously received EGFR monoclonal antibody therapy.
2. Have received anti-tumor treatments such as chemotherapy, biological therapy, targeted therapy, immunotherapy, etc. within 4 weeks prior to the first use of the study drug.
3. Have undergone major organ surgery (excluding biopsy) or experienced significant trauma within 4 weeks prior to the first use of the study drug.
4. Have received other clinical study drugs within 4 weeks prior to the first use of the study drug.
5. Known hypersensitivity or intolerance to any component of the study drug or its excipients.
6. Those who use strong or moderate CYP3A4 inducers within 14 days before the first administration of the study drug.
7. The adverse reactions of previous anti-tumor treatments have not yet recovered to CTCAE 5.0 evaluation ≤ level 1 except for toxicity such as alocepia, which is judged to be of no safety risk by researchers;
8. Central nervous system metastasis or meningeal metastasis with clinical symptoms.
9. Having a history of autoimmune diseases, immunodeficiency, including HIV testing positive, or having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.
10. Active hepatitis B (hepatitis B virus titer>1000 copies/mL or 200 IU/mL); Hepatitis C virus and syphilis infections.
11. Have a history of serious cardiovascular disease.
12. Unable to swallow medication orally, or has a condition that has been determined by researchers to seriously affect gastrointestinal absorption.
13. Within 5 years prior to the first use of the study drug, there were other malignant tumors, except for localized tumors such as cervical carcinoma in situ, basal cell carcinoma of the skin, and prostate carcinoma in situ that have been confirmed to be cured.
14. Any evidence of a history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, or clinically active interstitial lung disease.
15. Patients with a history of other serious systemic diseases who have been determined by the researchers to be unsuitable for clinical trials.
16. Known to have alcohol or drug dependence.
17. Has a clear history of neurological or psychiatric disorders, including epilepsy or dementia.
18. Pregnant or lactating women.
19. The researchers believe that the subjects are not suitable to participate in this clinical study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Adverse events incidence and severity | Up to approximately 60 months after the first participant was enrollment
Overall Response Rate（ORR）per RECST 1.1 | Up to approximately 60 months after the first participant was enrollment

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 60 months after the first participant was enrollment
Progression Free Survival (PFS) per RECIST 1.1 | Up to approximately 60 months after the first participant was enrollment
Duration of Response (DoR) per RECST 1.1 | Up to approximately 60 months after the first participant was enrollment
Disease Control Rate (DCR) per RECST 1.1 | Up to approximately 60 months after the first participant was enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Li Zhang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No